CLINICAL TRIAL: NCT03218228
Title: Evaluation of the Health of Peri-implant Tissues Around Immediately Placed Dental Implants in Aggressive Periodontitis Patients Versus Periodontally Healthy Individuals in Maxillary Esthetic Zone
Brief Title: Immediate Implant Placement in Aggressive Periodontitis
Acronym: implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nermin mohammed ahmed yussif, principal investigator-faculty of oral and dental medicine, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: immediate implant
Record Dates: First submitted 2017-07-03; First posted 2017-07-14 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Periodontitis
Keywords: aggressive periodontitis
MeSH Terms: conditions — Periodontitis; Aggressive Periodontitis | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implants in healthy individuals (Placebo Comparator): immediate placement of dental implants in individuals with healthy periodontium. the device is dental implants, radiographs, william's periodontal probe
  Interventions: Procedure: implants in periodontitis
- implants in periodontitis patients (Experimental): immediate implantation in patients suffering from aggressive periodontitis. the device is the dental implants, radiographs, william's periodontal probe
  Interventions: Procedure: implants in periodontitis

INTERVENTIONS:
Procedure: implants in periodontitis — it targets immediate implant placement in patients suffering from aggressive periodontitis
  Other Names: implants in aggressive periodontitis

SUMMARY:
The aim of the present study is to evaluate the health of immediately placed dental implants in aggressive periodontitis patients versus those placed in periodontally healthy individuals in the maxillary esthetic zone.

DETAILED DESCRIPTION:
Aggressive periodontitis is an enigmatic periodontal disease that characterized by massive and undeterminable periods of tissue destruction. It gets along well to young individuals with successive periods of disease activity. Aggressive bone destruction with limited plaque and calculus deposits usually detected. According to microbial theory, Aggregatibacter actinomycetemcomitans (A.a) and P. gingivalis (P. G) were claimed for such a disease. Patients of aggressive periodontitis have disturbed esthetic and masticatory function problems.

After wards, microbial theory was modified to enroll the genetic background that can be the cause behind the developed body resistance. Although the importance of the genetic treatment to improve the body response, it was totally dismissed during the routine periodontal work attributable to high cost effectiveness of the needed genetic analysis especially in developing countries.

Further researches tried to explain the cause behind the impaired body response. Impaired functions of the immune cells and the massive amounts of catabolic cytokines such as IL-1, IL-6, Il-17, TNF- α and prostaglan¬din E2 (PGE2) are usually released during the active periods of the disease. On the other hand, matrix-metalloproteinases are destructive enzymes that released in an uncontrollable manner. Host modulators were suggested to control the released of the destructive agents.

Immediate implant placement provides an efficient modality that shortens the dental management period. The aim behind immediate implant placement is the proper implant positioning to counteract the advanced bone resorption following extraction.

Periodontitis is considered an important risk factor for peri-implantitis. The pre-existing periodontitis must be treated prior to implant placement in order to avoid the bacterial accumulation in the periodontal lesions regardless the type of periodontitis. Local and systemic supportive therapy is strongly recommended in order to reduce the microbial colonies and post-operative bone loss.

Higher rate of implant failure (peri-implantitis) has been reported in immediately placed implants when compared with the delayed conventional technique. The failure rate markedly increased with the immediate placement of implants in patients with history of periodontitis especially the aggressive form.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects aged above 18 years old.

  * Patients should be free from any systemic disease.
  * patients with good oral hygiene
  * completely or partially edenthulus patients

Exclusion Criteria:

* Current and former smokers.

  * Pregnant females.
  * Patients with systemic diseases that may interfere with periodontal condition
  * Uncooperative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-10 (Actual); Primary Completion 2018-08-08 (Estimated); Study Completion 2018-12-08 (Estimated)

PRIMARY OUTCOMES:
implant and peri-implant tissues health | 12 months following implant placement
  it includes evaluation of the health of the placed implant in aggressive periodontitis patients and the surrounding alveolar bone and soft tissue. in other wards it evaluate the survival rate of the dental implants placed in aggressive periodontitis patients. the health condition of the placed implants are evaluated according to scale called health scale which include 5 categories in which probing depth, alveolar bone ressorption, mobility, pain and other items are measured).

SECONDARY OUTCOMES:
midfacial peri-implant mucosal level | 12 months following implant placement
  evaluattion of the mucosal level at the midfacial site of the immediately placed dental implants

CONTACTS AND LOCATIONS:
Overall Officials: mona darhous, Prof, Study Director — faculty of oral and dental medicine cairo university
Locations (1):
- Octobar University of Modern Sciences and Arts, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No